CLINICAL TRIAL: NCT07014579
Title: Utilizing LifeMap To Investigate Malignant Arrhythmia Therapeutic Efficacy in Athletes
Brief Title: Using Heart Electrical Signals to Study How Well Treatments Prevent Dangerous Heart Rhythms in Active People
Acronym: ULTIMATE-A
Status: Not yet recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 1037; NIHR203327 (Other Grant/Funding Number: National Institute for Health and Care Research Leicester Biomedical Research Centre)
Record Dates: First submitted 2025-05-28; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Inherited Cardiac Conditions; Sudden Cardiac Arrest; Ventricular Arrhythmia; Athlete; Ventricular Fibrillation
Keywords: ULTIMATE-Athlete; LifeMap; R2I2; PERS; Ventricular Arrhythmia; Ventricular Fibrillation; Sudden Cardiac Death
MeSH Terms: conditions — Death, Sudden, Cardiac; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants with ICD: Those that exercise 3 hours or more per week and/or have a physically active occupation (e.g military, fire service, landscaper, etc.) and have been identified as at risk of sudden cardiac death. Therefore have been implanted with an implantable defibrillator (ICD) for primary or secondary prevention.
- Participants without heart device: Those that exercise 3 hours or more per week and/or have a physically active occupation (e.g military, fire service, landscaper, etc.) and do not have any heart condition. Therefore have not been implanted with any heart device.
- Participants with Pacemaker: Those that exercise 3 hours or more per week and/or have a physically active occupation (e.g military, fire service, landscaper, etc.) and have not been identified as at risk of sudden cardiac death. Therefore do not have an implantable cardioverter defibrillator, but have been implanted with a cardiac pacemaker due to other conditions.

SUMMARY:
The goal of this observational study is to learn if two specific heart electrical signal patterns can help in detecting the risk of dangerous heart rhythms in athletes, and to see if exercise-based tests can be used instead of invasive hospital procedures to record this electrical signals.

The main questions it aims to answer are:

1. Can special ECG action potential duration markers (R2I2 and PERS) identify athletes who are at higher risk of sudden heart rhythm problems.
2. Can an exercise test give the same information as a non-invasive electrophysiology study.

Researchers will compare athletes who have an implanted heart device (ICD) with athletes who do not, to see if there are differences in these heart signals.

Participants will undergo:

1. ECG recordings during rest and exercise.
2. If they have an ICD or pacemaker, an ECG will be recorded during a non invasive stimulation.
3. A continuous 24 hour ECG.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over.
* Participates in regular physical activity for at least 3 hours or greater weekly.
* Having Implantable cardioverter defibrillator insitu (cases).
* Having a cardiac pacemaker (control).
* Having no cardiac device (control).
* Sufficient capacity and agreement to participate orally and signed written consent forms.
* Understanding of written and spoken English language.

Exclusion Criteria:

* Pregnancy, as detected by positive urine pregnancy test result.
* Inability to comply with study protocols.
* Any iatrogenic cardiac pathology (stents, CABG etc).
* Unstable ventricular tachycardia (>30 seconds).
* Any unstable malignant arrhythmia.
* Fever or presence of a clinically diagnosed febrile illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be from a single tertiary care hospital (University Hospitals Leicester), and residents of United Kingdom
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Restitution Markers as Determined by R2I2 and PERS | The primary outcome measure is assessment of changes in the regional restitution instability index and peak ECG restitution slope at various time points including, baseline, during 15-minute exercise and during 15-minute electrophysiology study.

SECONDARY OUTCOMES:
Non-invasive exercise-based tests correlate with electrophysiology study. | The secondary outcome looks at how the Regional Restitution Instability Index (R2I2) and Peak ECG restitution slope (PERS) measurements during a 15-minute exercise compare with those taken during 15 minute Non-Invasive Programmed Stimulation (NIPS).

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam André Ng, MBChB, MRCP, Ph.D, FRCP, Study Director — University of Leicester, Leicestershire, United Kingdom; Ghulam André Ng, MBChB, MRCP, Ph.D, FRCP, FHEA, Principal Investigator — University of Leicester, Leicestershire, United Kingdom; Xin Li, PhD, MSc, BSc, FHEA, Principal Investigator — University of Leicester, Leicestershire, United Kingdom; Harshil Dhutia, MBBS, BSC, MRCP, CCDS, MD(RES), Principal Investigator — Glenfield Hospital, Leicester
Locations (1):
- Glenfield Hospital, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet due to study committee and study sponsor needing to deliberate

REFERENCES:
- [Background] Nicolson WB, Smith MI, Vali Z, Samani NJ, Ng GA. Application of two novel electrical restitution-based ECG markers of ventricular arrhythmia to patients with nonischemic cardiomyopathy. Pacing Clin Electrophysiol. 2021 Feb;44(2):284-292. doi: 10.1111/pace.14143. Epub 2021 Jan 4. PMID 33336815
- [Background] Ng GA, Mistry A, Li X, Schlindwein FS, Nicolson WB. LifeMap: towards the development of a new technology in sudden cardiac death risk stratification for clinical use. Europace. 2018 Sep 1;20(FI2):f162-f170. doi: 10.1093/europace/euy080. PMID 29684162
- See also: LifeMap is a novel, highly promising technique for assessing risk of sudden cardiac death, a condition that kills 3 million people annually — https://life-map.co.uk/